CLINICAL TRIAL: NCT06378736
Title: Test of Whether Theta-gamma Coupling Present in Electroencephalogram Recording in Patients With Systemic Lupus Erythematosus Acts as an Objective Marker for Cognitive Dysfunction
Brief Title: Electroencephalogram Recording in Patients With Systemic Lupus Erythematosus
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Bruce Volpe, Professor, Investigator, Northwell Health
Other Study IDs: 21-1027
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (5 ml) will be drawn and processed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Electroencephalography (EEG) signals, which will be detected noninvasively from dry scalp surface electrodes while the subjects are in a state of wakeful rest. — The proposed study is to determine whether EEG signals, namely theta-gamma coupling (TGC); The investigators are testing whether TGC can be used as a non-invasive novel biomarker in diagnosis and monitoring of insidious and difficult to detect cognitive dysfunction in SLE patients.

SUMMARY:
Patients with systemic lupus erythematosus (SLE) often experience a frustrating decline of their cognitive skills that includes considerable problems in attention, learning, and memory. This lupus-related cognitive dysfunction (termed SLE-CD) is recognized as the most prevalent of the nineteen neuropsychiatric SLE syndromes, as it affects up to 80% of patients and can significantly decrease their quality of life. The goal is to have tools that can be used for diagnosis and for monitoring responses after targeted interventions and therapies. This study will focus on electroencephalographic (EEG) signals, which will be detected noninvasively from scalp placed surface electrodes while the subjects are in a state of wakeful rest. Our hypothesis is that a subset of brain oscillations known as theta and gamma, and their co-modulation or coupling will be disrupted in SLE patients. This research protocol will subject patients with systemic lupus erythematosus (SLE) to scalp electroencephalography (EEG), with the goal of determining whether specific EEG patterns ('theta-gamma coupling') appear abnormal during wakeful-rest periods of 20 minutes. The investigators are interested in using scalp EEG because it is a standard, safe and robust technique for monitoring the electrophysiological activity of neurons in the cerebral cortex.

DETAILED DESCRIPTION:
Patients will sit comfortably in a quiet room in a wakeful state and perform simple operations with toy blocks and look at three dimensional objects and answer some questions. The EEG electrodes fit into a custom-made cap and will effectively transmit wave activity just by touching the skin surface of the scalp. There is no need for electrode paste so at the end of the experiment the patient can remove the cap and go home. The entire procedure including fitting of the EEG cap will take about an hour.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and provide informed consent.
2. Must be ≥18 and ≤65years of age.
3. Must be female.
4. Must fulfill the 1997 American College of Rheumatology (ACR) revised criteria for the diagnosis of SLE or the Systemic Lupus Erythematosus International Collaborating Clinics (SLICC) Criteria for SLE.
5. Must have stable disease activity and medication doses for 4 weeks prior to screening. Stable disease activity is defined as no increase in disease activity requiring an increase or change in medications.
6. Must be on a corticosteroid dose that is ≤ prednisone 10 mg daily, or equivalent.
7. Aim 1 ONLY: Must have demonstrated significantly increased metabolism in the hippocampus, temporal or parietal lobes on prior fluoro-deoxy glucose (FDG)-PET imaging.

Exclusion Criteria:

1. Inability or unwillingness to give written informed consent or comply with study protocol.
2. History of neurological diseases including, but not limited to, severe head injury or history of brain surgery, stroke, seizure, toxic exposure, mental retardation, migraine headaches, multiple sclerosis, dementia.
3. History of documented transient ischemic attacks within 6 months of screening.
4. History of illicit drug or alcohol dependence/abuse within the past 12 months.
5. Current use of antipsychotic, anticonvulsant, antidepressant (except for selective serotonin reuptake inhibitors) or anxiolytic medications (short acting anxiolytic medications are allowed if taken as needed with > 5 half-lives prior to assessments).
6. History of chronic pain; current and/or chronic use of narcotic analgesia for > 21 days (total) within the last 3 months, or last dose less than 5 days prior to assessment.
7. Increased disease activity within 4 weeks of screening defined by an increase in SLEDAI by 3 points or more, exclusive of points from serologies, which prompts an increase in or new addition of SLE medications.
8. History of a diagnosis of a primary psychiatric disorder preceding SLE diagnosis.
9. Current active acute infections requiring antibiotics within 2 weeks of screening and chronic known infections (eg. hepatitis B, C, and/or HIV).
10. Co-existing other autoimmune disease(s) other than autoimmune thyroid disease and secondary Sjogren's Syndrome.
11. The presence of uncontrolled, severe hypertension, diabetes or heart disease.
12. Impaired renal function with an estimated glomerular filtration rate (eGFR)< 30.
13. Presence of any active medical condition that in the opinion of the investigator may contribute to cognitive and/or behavioral disturbances.
14. Use of investigational drugs within 30 days or 5 half-lives before the study visit, whichever is longer.
15. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
16. Current treatment with cyclophosphamide, addition of belimumab within 4 months, addition of any disease modifying drug or biologic within 3 months of screening, and/or rituxan within 6 months.
17. Limited fluency with English or Spanish that in the opinion of the investigator would limit the subject's performance on the assessments.
18. Pregnant and/or lactating women.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Twenty of the SLE subjects that have participated in prior brain imaging studies. The other 20 SLE subjects will be recruited from 2 ongoing observational studies of brain involvement in SLE.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
A measure of the amount and relationship of theta and gamma waves in the EEG recording. The ability to perform the block building task and the ability to choose among unfolded three-dimensional objects. | Aim 1 will take the first 24 patients and they will spend an hour and a half undergoing EEG measuring TGC. For Aim 2 the patients will undergo EEG measuring TGC and predict the subsequent PET scan - which will occur under a separate protocol.
  Patient will build with toy blocks and three dimensional combination will suffice. The patient will also observe three dimensional objects - cubes, for example, that are unfolded and choose a matching object from an array that includes the object and three foils. EEG activity will be recorded during this period.
  As the subjects will be fitted with noninvasive EEG caps (using dry electrodes that will contact the scalp directly) which will record the ongoing brain activity while the subjects, in a wakeful resting mode attempt to build with the toy blocks and analyze the three dimensional figures. This activity will go on for approximately 20 minutes.
  The EEG signals will be analyzed to determine the theta gamma coupling (TGC).

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health-Feinstein Insitute, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make recordings available to qualified researchers and pay attention to keep protected health information (PHI) confidential.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the complete analysis of the patient groups and after complete analysis of the healthy control group.
Access Criteria: To be determined.